CLINICAL TRIAL: NCT03218722
Title: Impact of Early Administration of Prothrombin Concentrate Complex in Patients With Acute Hemorrhage Following Severe Trauma
Brief Title: Early Administration of Prothrombin Concentrate Complex in Patients With Acute Hemorrhage Following Severe Trauma
Acronym: PROCOAG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 38RC16.046
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Shock, Hemorrhagic
Keywords: Acute traumatic coagulopathy; Hemostasis; Severe hemorrhage
MeSH Terms: conditions — Shock, Hemorrhagic; Hemorrhage | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCC treatment (Experimental): Conventional strategy for ATC management in addition to of intravenous Pro-Thrombin Concentrate Complex (25IU/kg factor IX)
  Interventions: Drug: Pro-Thrombin Concentrate Complex
- Placebo treatment (Placebo Comparator): Conventional strategy for ATC management without PCC (NaCl 0.9%)
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Pro-Thrombin Concentrate Complex — Patient at risk of massive hemorrhage will be managed with standard care with 1ml/kg PCC.
  Other Names: KANOKAD
  Arms: PCC treatment
Drug: NaCl 0.9% — Patient at risk of massive hemorrhage will be managed with standard care with 1ml/kg Saline solution.
  Arms: Placebo treatment

SUMMARY:
Acute traumatic coagulopathy (ATC) is common in severe trauma patients (around 25 to 30% of patients with severe trauma) and is associated with increased mortality. ATC is associated with fibrinogen and clotting factors deficiencies. Therefore, ATC management relies on early administration of fibrinogen and blood products in case of massive transfusion with a 1:1 or 1:2 ratio between Fresh Frozen Plasma (FFP) and Red Blood Cells (RBC). This strategy relies on fast supply of FFP.

To overcome delay for FFP ordering, transport and defrosting, the PROCOAG study proposes to use prothrombrin concentrate complex (PCC) as alternative to treat coagulation factor deficiency. PCC is readily available upon hospital arrival. In addition to fibrinogen treatment, it is thought that PCC can be efficient in ATC management, while reducing risks associated with massive transfusion.

ProCoag is a randomized, controlled, double-blinded, parallel clinical trial aiming at showing superiority of early PPC+ fibrinogen strategy on fibrinogen only strategy for the management of patients at risk of massive transfusion.

Early administration of PPC should optimize patient blood management and therefore reduce blood products transfused within the first 24 hours following a severe trauma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary admission for a severe trauma
* Out-of-hospital transfusion or RBC transfusion within the first hour following hospital admission
* Clinical prediction or ABC score (Assessment of Blood Consumption) ≥ 2 of massive transfusion defined by a transfusion of at least 10 CGR during the first 24 hours or 3 CGR during the first hour.
* Informed consent signed by a relative or emergency procedure

Exclusion Criteria:

* Cardiac arrest before randomisation
* Secondary transfer from another hospital (a technical stop is accepted)
* Post-traumatic lesions out of therapeutic resources with death expected in the hour following hospital admission
* Anti-coagulation treatment (K anti-vitamine, new oral anticoagulant)
* Pregnancy
* Hypersensitivity to active substances or one of the excipients of KANOKAD®
* Patient treated with an experimental medicine within the last 30 days
* Decision of therapeutic limitation before randomisation
* Patient protected by article L1121-7 of the French Public health code.
* Knowledge of a contraindication to the use of NaCl 0.9% at the dose of 1 mg/kg (hyperchloremia, hypernatremia...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Labile blood products transfused in the first 24 hours | 24 hours following hospital admission
  This outcome is measured in number of bags administered

SECONDARY OUTCOMES:
RBC (Red Blood Cells) transfused in the first 24 hours | 24 hours following hospital admission
  This outcome is measured in number of bags administered
FFP transfused in the first 24 hours | 24 hours following hospital admission
  This outcome is measured in number of bags administered
Platelets transfused in the first 24 hours | 24 hours following hospital admission
  This outcome is measured in number of bags administered
Time to achieve Prothrombin ratio < 1.5 | Within the first 24 hours
Time to hemostasis | Within the first 24 hours following admission
  Hemostasis is defined as bleeding control in the surgical field or resolution of contrast blush after embolization during interventional radiology
Thrombo-embolic events | ICU stay (an average of 28 days)
Mortality | 24 hours and Day 28
ICU-free days | Hospital stay (an average of 28 days)
  Number of in-hospital days outside Intensive Care Unit (ICU)
Ventilator-Free Days | ICU stay (an average of 21 days)
  Number of days without mechanical ventilation
Hospital-free days | Within the first 28 days
  Number of days outside hospital
Glasgow Outcome Scale Extended (GOSE) | Day 28
Hospitalisation status | Day 28
Cost of the strategy | Day 8 and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOUZAT, Principal Investigator — CHU Grenoble Alpes
Locations (12):
- France (12):
  - Annecy University Hospital, Annecy
  - AP-HP Beaujon, Clichy
  - Grenoble University Hospital, Grenoble
  - AP-HP Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Lille University Hospital, Lille
  - HCL - Hôpital Edouard Herriot, Lyon
  - AP-HM - Marseille Nord, Marseille
  - Montpellier University Hospital, Montpellier
  - Nantes University Hospital, Nantes
  - AP-HP Pitié Salpetrière, Paris
  - HCL - Lyon Sud, Pierre-Bénite
  - Strasbourg University Hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouzat P, Charbit J, Abback PS, Huet-Garrigue D, Delhaye N, Leone M, Marcotte G, David JS, Levrat A, Asehnoune K, Pottecher J, Duranteau J, Courvalin E, Adolle A, Sourd D, Bosson JL, Riou B, Gauss T, Payen JF; PROCOAG Study Group. Efficacy and Safety of Early Administration of 4-Factor Prothrombin Complex Concentrate in Patients With Trauma at Risk of Massive Transfusion: The PROCOAG Randomized Clinical Trial. JAMA. 2023 Apr 25;329(16):1367-1375. doi: 10.1001/jama.2023.4080. PMID 36942533
- [Derived] Bouzat P, Bosson JL, David JS, Riou B, Duranteau J, Payen JF; PROCOAG study group. Four-factor prothrombin complex concentrate to reduce allogenic blood product transfusion in patients with major trauma, the PROCOAG trial: study protocol for a randomized multicenter double-blind superiority study. Trials. 2021 Sep 16;22(1):634. doi: 10.1186/s13063-021-05524-x. PMID 34530886